CLINICAL TRIAL: NCT02637674
Title: Uterine Allotransplantations Using Uterine Grafts From Brain-dead Female Donors
Acronym: ATU
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I14002/ATU
Record Dates: First submitted 2015-12-10; First posted 2015-12-22 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Infertility
Keywords: allotransplantation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Uterus Transplantation (Experimental): Women will undergo deceased donor uterine transplantation after IVF
  Interventions: Procedure: Uterus Transplant

INTERVENTIONS:
Procedure: Uterus Transplant

SUMMARY:
Uterus transplantation may enable women with uterine factor infertility to become pregnant and give birth.

This study will explore the feasibility of a uterine transplant and eight subjects will undergo deceased donor uterine transplantation at CHU de Limoges.

There phases involved in this study: Primary, Secondary and Tertiary Screening, Medical Evaluation, IVF, Transplantation, Embryo Transfer, Pregnancy/Delivery and Follow up.

DETAILED DESCRIPTION:
It is estimated that 1 in 500 women of reproductive age have congenital or acquired uterine factor infertility (UFI).

The solution for such patients who wish to have a child is either to adopt or use a surrogate. The latter is illegal in France .Uterine transplantation (UT) could be a beneficial medical alternative.

Over the last 13 years, about 30 experimental studies have been conducted on rodents, rabbits, pigs, sheeps and monkeys. They have shown TU to be feasible, with a number of births achieved after uterus auto-transplantation, syngeneic transplantation and allotransplantation. However, animal experiments are not able to provide a definitive answer to the question of the feasibility of UT in women due to the specific characteristics of each species and a lower degree of control of immunosuppression and in vitro fertilisation techniques in animals. Thus, the information from animal experiments and the present knowledge on immunosuppression in women, based on experiments in other solid organ transplantation, explain the willingness to take the step of undergoing clinical UT. The recent human data and the first births after UT obtained by a Swedish team are reassuring and confirmed the feasibility of the procedure. The data gathered over 50 years of pregnancies in patients who have received kidney, liver or heart transplants is reassuring, with over 20,000 births recorded and recommendations for the start of the pregnancy, patient follow-up and immunosuppressive drugs (ISD) handling are currently relatively well-established.

As compared to other solid organ transplantations, UT is particular in being temporary (the graft will be removed once the child is born or in case of safety issue) and the period of exposure to immunosuppressants is thus reduced.

Our team has recognised experience in the field of female fertility preservation and ovarian grafting. Work begun in animals at the end of the 1990s led to the first pregnancies in France after an ovarian autograft in 2010. With regard to uterus grafting, the investigators have published work on uterine allotransplantation involving ewes and the evaluation of the graft by magnetic resonance imaging (MRI). Clinically, the investigator began by working on cadavers and conducted a study in 2012-2013, which was supported by the French Biomedical Agency (Agence de la biomédecine), on the feasibility of uterus retrieving as part of a multi-organ retrieval (MOR) procedure. In this preliminary clinical study, the investigators were able to show that the technique of uterus retrieval in brain-dead donors can be reproduced. Acceptance of the retrieval by the relatives of the brain-dead patient was good (no refusal).

In the present protocol, the investigators propose a pilot study of UT in women with grafts from brain-dead female donors.

In humans, UT can be envisaged with grafts from either living or deceased donors. In Turkey, a UT with a brain-dead donor, performed in 2011, was the first to achieve a pregnancy. This pregnancy was, unfortunately, non-progressive. In Sweden, the team of Prof. Brannström performed nine UTs in 2012 and 2013 with living donors. One donor suffered a utero-vaginal fistula, thus confirming the potential surgical risk of such a procedure for living donors. Conversely, for the recipients, the success rate of UT after six months was 78% (seven successful transplantations, with a menstrual period occurring in the first six months, out of the nine transplantations performed).

Unlike the Swedish team, the investigators are planning to use grafts from brain-dead donors in order to avoid the potential surgical risks with alive donors. In addition, according to the French Biomedical Agency, there are around 220 brain-dead female donors below 50 years each year in France.

The recipients will be selected according to the inclusion criteria. They will be asked to promise to live close to Limoges University Hospital during the 3 months post uterus transplantation. Inclusion will be confirmed if none of the primary, secondary or tertiary exclusion criteria is present and if at least 10 embryos are obtained via IVF conducted at Limoges University Hospital. The patients will then be registered on a transplant waiting list. Since the aim of the project is to perform eight UTs, any patient who has signed the consent form can be replaced if she is secondarily excluded or wishes to withdraw from the study.

The uterine retrievals will be performed by the surgical team of Limoges University Hospital in four retrieval centres in the central-western part of France.

Uterine transplantation will be performed in Limoges University Hospital by the vascular and gynaecological surgery teams. Patients will then be monitored jointly by the gynaecology, renal transplantation and psychiatric teams. The immunosuppressive treatment will include an induction (anti-CD25 antibodies), tacrolimus, antimetabolites (mycophenolate mofetil followed by azathioprine before and during pregnancy) and an initial corticotherapy. The graft will be monitored by imaging (MRI, ultrasound), biopsy of the cervix and therapeutic drug monitoring. Rejection will be determined according to the criteria of Johannesson.

The success of transplantation will be confirmed by the occurrence of a menstrual period during the first year.

In successful cases, embryo transfers will begin on the second year of transplantation. In the absence of a successful pregnancy, the transfer attempts will continue each month until there are no available embryos left, and for a maximum period of 18 months. The embryos that have not been used will be managed in accordance with the French law on bioethics. The patient will receive close multidisciplinary follow-up throughout the pregnancy. The delivery will be done by caesarean section. The graft will be explanted immediately following the caesarean when possible or 2 months post partum.

If the UT fails (no menstrual period in one year), the graft will be explanted. The graft will also be explanted in the following situations: uterine necrosis, corticoresistant rejection, serious adverse effects attributable to immunosuppressive drugs, severe infectious complications, haemorrhagic complications, the absence of a progressive pregnancy after a maximum period of 18 months of embryo transfer attempts, separation of the couple.

The children will receive follow-up from a paediatrician in accordance with common practice. All live attenuated vaccines will be contraindicated in the first six months following birth.

ELIGIBILITY:
Inclusion Criteria:

Recipients :

Primary selection criteria

Patients with uterine factor infertility defined as followed :

* A history of hysterectomy for benign pathology or postpartum haemorrhage
* Total or partial uterine agenesis

  * Age ≥ 25 and < 35 years
  * couple living together for at least two years
  * BMI ≤ 30 kg/m2
  * At least 12 months from colpoplasty surgery
  * At least 12 months from diagnosis of uterine infertility
  * Nulliparous
  * Compliance with the legal criteria of medically assisted procreation Acceptance to take part of NEHAVI cohort
  * Acceptance of the protocol constraints
  * Coverage by the French national Health service

Secondary selection criteria

* Signed informed consent by the patient and spouse
* Prior psychological evaluation not contraindicating participation in the study
* Normal ovarian function and satisfactory ovarian reserve
* Compliance with primary selection criteria.

Tertiary selection criteria

* At least 10 embryos obtained by IVF
* Compliance with primary and secondary selection criteria

Donors

• Brain dead female ≥ 18 years old and ≤ 50 years old.

Exclusion Criteria:

Recipients Primary criteria for non-selection

* • Previous major abdomino-pelvic surgery
* Previous ileal or sigmoid colpoplasty
* History of cancer
* Active tobacco consumption
* Hypertension (HT), including treated HT
* Type 1 or 2 diabetes
* Chronic kidney disease
* Evolving cardiovascular pathology
* Psychiatric disease
* Under guardianship or conservatorship
* Contraindication to one of the treatments used in the study
* Contraindication to ovarian stimulation treatment except uterine infertility

Secondary criteria for non-selection

* Prior psychological evaluation contraindicating participation in the study
* Rare blood group AB or B, for the purpose of reducing the waiting time for a graft. Groups A and O combined constitute over 85% of donors (see appendix)
* Positive irregular agglutinin test (IAT)
* Ovarian insufficiency according to laboratory norms
* Presence of anti-HLA antibodies
* Negative Epstein-Barr virus serology
* HIV or hepatitis C infection,
* Hepatitis B (acute, chronic, treated)
* Presence of a single kidney
* Detected cardiac pathology
* Contraindication to participation into the trial detected at the anaesthetic assessment
* Dermatological, stomatological and/or ear, nose, and throat (ENT) pathology/ies contraindicating treatment with ISDs
* Thoracic-abdominal-pelvic CT scan anomalies contraindicating UT and the use of treatment with ISDs
* Increased risk of miscarriage (thrombophilia, anormal karyotype)
* Separation of the couple.

Tertiary criteria for non-selection

* Spouse/partner with azoospermia
* Less than 10 frozen embryos obtained
* Separation of the couple.
* Previous uterine transplantation

Donors

* Length of no flow > 10 min
* Pregnancy at the time of brain death
* Time from delivery < 3 months
* Positive oncogen human papillomavirus (HPV )test (16 and 18)
* Myomas > 3 cm and/or endoluminal fibroid and/or endometrial polyps and/or heterogenous annexial cyst seen in a pelvic ultrasound or CT scan
* Multi-scarred uterus ( ≥ 2 uterine scars)
* Registered in the national registry of persons who refuse to donate any organ.
* Opposition to the uterine retrieval from the donor's relatives.
* Uterine agenesis and uterine malformation
* Criteria usually seen as contraindicating retrieval (HIV+, evolutive neoplasia, etc.)

Ages: 25 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Successful uterus transplant | 12 month after each transplantation
  Success will be measured by by the occurrence of at least two spontaneous menstrual cycles during the first year following the UT.

SECONDARY OUTCOMES:
UT complications | up to 41 after transplantation
Successful of pregnancies achieved | up to 30 months after transplantation
Pregnancy complications after UT | up to 39 months after transplantation
Successful of births achieved | up to 39 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Tristan GAUTHIER, Doctor, Principal Investigator — University Hospital, Limoges
Locations (4):
- France (4):
  - Service de gynécologie, Limoges
  - Service de néphrologie, Limoges
  - Service de Pharmacologie, Limoges
  - Service de réanimation, Limoges